CLINICAL TRIAL: NCT00669175
Title: Safety and Efficacy of a Low Dose Naloxone Infusion in NICU Patients
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Eugenia Pallotto, Children's Mercy Hospital
Other Study IDs: 08 01-003
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Opioid Tolerance; Pain
Keywords: Naloxone; Neonate; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
When narcotic pain medicine, like fentanyl or morphine, is given to adults and children for several days, they often develop a tolerance to the medicine. This means they may need higher doses over time to get the same amount of pain control. When it is time to stop the medicine, the dose has to be decreased slowly so that the patient does not have withdrawal symptoms.

Naloxone is a medicine that at high doses can reverse the effects of narcotics. At very small doses it may help prevent tolerance and lessen the severity of withdrawal symptoms. This could mean less narcotic pain medicine is needed over fewer days.

The purpose of this research study is to see if giving naloxone to neonates who require narcotic infusions is safe and effective. Safety will be measured by the incidence of side effects. Efficacy will be measured by monitoring for changes in pain and sedation scores and need for more pain medicine.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single center, open label dose escalation study. We hypothesize that critically ill patients in the NICU may benefit from a low dose naloxone infusion resulting in decreased tolerance, less severe withdrawal symptoms, lower cumulative doses of opiates, and fewer total days of opiates, all while maintaining adequate or enhanced pain control and sedation. Establishing safety and efficacy data for this potentially beneficial therapy is an important first step towards using this therapy to decrease the risk of opioid tolerance and withdrawal in this population of infants.

ELIGIBILITY:
Inclusion Criteria:

* Neonates > 36 0/7 weeks estimated gestational age
* Less than 30 days of life
* Requiring admission to to the Neonatal Intensive Care Unit
* Requiring continuous infusions of fentanyl or morphine analgesia
* Anticipated to require opioid infusions for at least four days
* Patients must be enrolled within 120 hours of initiating opioid infusions
* All patients will also require mechanical ventilation prior to study entry.

Exclusion Criteria:

* Preterm infants < 36 weeks gestation
* Neonates with major neurologic anomalies, seizures
* Opioid infusion administration for > 120 hours prior to study entry
* Patients requiring ECMO support prior to study entry
* Neonates born to mothers who are known to be opioid dependent

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates admitted to the NICU within the first five days of life with an anticipated need for opiate infusion for at least four days
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-02; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be a change in N-PASS scores. N-PASS scores will be compared before, during, and after administration of naloxone. | Before, during, and after administration of naloxone

SECONDARY OUTCOMES:
The secondary outcome variable will be any changes in dosing of opioids within four hours of initiating or increasing naloxone infusion. Vital signs will be recorded per NICU protocol and closely monitored for changes. | Collected and compared for the time period before, during, and for 5 days after naloxone infusion is administered

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia K Pallotto, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States